CLINICAL TRIAL: NCT04016077
Title: A PHASE 1, NON-RANDOMIZED, OPEN LABEL, MULTIPLE DOSE STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF 06651600 IN SUBJECTS WITH HEPATIC IMPAIRMENT AND IN HEALTHY SUBJECTS WITH NORMAL HEPATIC FUNCTION
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of PF-06651600 in Subjects With Hepatic Impairment and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B7981016
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Hepatic Impairment; Healthy Participants
Keywords: PF-06651600; Pharmacokinetics; Hepatic impairment
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-06651600 Moderate Hepatic Impairment (Experimental): This arm includes participants with moderate hepatic impairment who will receive oral doses of PF-06651600 30 mg on Day 1 through Day 10.
  Interventions: Drug: PF-06651600 30 mg
- PF-06651600 Healthy participants (Experimental): This arm includes healthy adult participants who will receive oral doses of PF-06651600 30 mg on Day 1 through Day 10.
  Interventions: Drug: PF-06651600 30 mg
- PF-06651600 Mild Hepatic Impairment (Experimental): This arm is in Part 2 which will be conducted if the decision criterion to proceed to Part 2 is met.
  The arm includes participants with mild hepatic impairment who will receive oral doses of PF-06651600 30 mg on Day 1 through Day 10.
  Interventions: Drug: PF-06651600 30 mg

INTERVENTIONS:
Drug: PF-06651600 30 mg — PF-06651600 in 10 mg oral tablets will be administered on days 1 to 10.

SUMMARY:
The purpose of this study is to characterize the effect of hepatic impairment on the pharmacokinetic(s) (PK) of PF-06651600 following administration of multiple once daily doses of PF-06651600. The safety and tolerability of PF-06651600 will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations and other study procedures
* Body mass index (BMI) of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lb)

Additional Inclusion Criteria for Participants with Normal Hepatic Function:

* Healthy male or female participants
* No known or suspected hepatic disease

Additional Inclusion Criteria for Participants with Impaired Hepatic Function:

* Stable hepatic impairment, defined as no clinically significant change in disease status within the last 30 days prior to the Screening visit
* No other ongoing clinically significant abnormalities based on medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory tests except for the abnormal findings that are related to the participant's hepatic impairment.
* Satisfy the criteria for Class A or Class B of the Child-Pugh classification (mild: Child-Pugh Scores 5-6 points, and moderate: Child Pugh Scores 7-9 points), within 28 days of investigational product administration.

Exclusion Criteria:

* Has active acute or chronic infection requiring treatment or history of systemic infection requiring hospitalization, incl. herpes zoster, herpes simplex, tuberculosis
* Infection with hepatitis B, hepatitis C or HIV
* Any condition affecting drug absorption, distribution, metabolism and excretion (eg, status post porta-caval shunt surgery, prior bariatric surgery, gastrectomy, ileal resection)
* Has malignancy, lymphoproliferative disorder, surgery or other condition not allowed per protocol

Additional Exclusion Criteria for Participants with Normal Hepatic Function:

- Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, gynecologic or allergic disease

Additional Exclusion Criteria for Participants with Impaired Hepatic Function:

- Has encephalopathy, severe ascites and/or pleural effusion, Child-Pugh score >9 or medical conditions (like hepatorenal syndrome, gastrointestinal hemorrhage, etc.) excluded per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Purohit V, Huh Y, Wojciechowski J, Plotka A, Salts S, Antinew J, Dimitrova A, Nicholas T. Leveraging Prior Healthy Participant Pharmacokinetic Data to Evaluate the Impact of Renal and Hepatic Impairment on Ritlecitinib Pharmacokinetics. AAPS J. 2023 Mar 28;25(3):32. doi: 10.1208/s12248-023-00792-8. PMID 36977960
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981016

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight participants were originally enrolled in each cohort. Two participants in moderate hepatic impairment cohort who discontinued from study treatment were included as "completed" and 2 additional participants were enrolled to ensure an adequate number of evaluable participants.
Groups:
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment were administered PF-06651600 30 milligram (mg) once daily (QD) for 10 treatment days.
- Normal Hepatic Function: Participants with normal hepatic function were administered PF-06651600 30 milligram (mg) once daily (QD) for 10 treatment days.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 18 participants who were included in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (6.88) | 57.4 (6.48) | 58.3 (6.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to 24 Hours (AUC24) for PF-06651600
Description: AUC24 of PF-06651600 pre and post dose.
Time Frame: Hour 0 (pre-dose) on Days 7, 8 and 9, and hour 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24 hours post-dose on Day 10
Population: The analysis population was defined as all participants treated who have at least 1 of the pharmacokinetic (PK) parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
nanogram*hour per milliliter (ng*hr/mL) | 454.5 (45) | 383.6 (16)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Geometric Means = 118.50, 90% CI 2-sided [87.96 to 159.64]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for PF-06651600
Description: Cmax is maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: The analysis population was defined as all participants treated who have at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
nanogram per milliliter (ng/mL) | 194.3 (49) | 186.9 (24)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Geometric Means = 104.00, 90% CI 2-sided [74.48 to 145.23]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) (All Causalities and Treatment-related)
Description: AEs with all causalities were any untoward medical occurrences in a study participant administered a product which did not necessarily had causal relationship with the treatment or usage. An SAE was an AE resulting in any of the following endpoints or deemed significant for any other reason: death; life threatening (immediate risk of death); inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; or considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline (Day 0) up to 28 days after last dose of study medication (Day 39)
Population: All participants assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 10 | 8
Participants
  AEs (all causalities) | 4 | 2
  AEs (treatment related) | 4 | 1
  SAEs (all causalities) | 1 | 0
  SAEs (treatment related) | 1 | 0

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, erythrocytes, leukocytes, neutrophils, prothrombin time, prothrombin intl. normalized ratio), chemistry (bilirubin, direct bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, albumin, sodium, potassium, calcium, bicarbonate and glucose), urinalysis (glucose, ketones, protein, hemoglobin, urobilinogen, bilirubin and nitrite). Each parameter was evaluated against commonly used and widely accepted criteria.
Time Frame: Baseline (Day 0) up to 28 days after last dose of study medication (Day 39)
Population: All participants assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 10 | 8
Participants | 9 | 2

5. Secondary Outcome: Number of Participants With Out of Range Vital Signs
Description: Vital signs included supine blood pressure, pulse rate and temperature. The pre-specified out of range criterion for supine diastolic blood pressure was change from baseline equal to or over than (≥) 20 millimeter of mercury (mmHg). Clinical significance of vital signs and out of range criterion were determined at the investigator's discretion.
Time Frame: Baseline (Day 0) up to 28 days after last dose of study medication (Day 39)
Population: All participants assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 10 | 8
Participants | 1 | 0

6. Secondary Outcome: Number of Adverse Events Leading to Discontinuation
Description: Adverse events result in participants discontinuations from the study drug.
Time Frame: Baseline (Day 0) up to 28 days after last dose of study medication (Day 39)
Population: All participants assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Number; unit: adverse events
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 10 | 8
adverse events | 2 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) up to Day 39 (28 days after last dose of study medication).
Description: Participants were only counted once per hepatic function group per event. If a participant had more than one occurrence in the same Preferred Term event category, only the most severe occurrence was counted.
Arm/Group | Moderate Hepatic Impairment | Normal Hepatic Function
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/8
Other Adverse Events (participants affected / at risk) | 3/10 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Impairment (N=10) | Normal Hepatic Function (N=8)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Impairment (N=10) | Normal Hepatic Function (N=8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT04016077/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT04016077/SAP_001.pdf